CLINICAL TRIAL: NCT05655624
Title: Effects of Pursed Lip Breathing With and Without Mat Pilates Training on Dyspnea, Physical Health and Thoracoabdominal Expansion in Obese Women
Brief Title: Effects of Pursed Lip Breathing With and Without Mat Pilates Training in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0319
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Obese Women
Keywords: Borg's scale; Dyspnea; IPAQ; Mat Pilates; obese women; Thoracoabdominal expansion
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Pursed lip Breathing along Mat Pilates Training
  Interventions: Other: Pursed lip Breathing along Mat Pilates
- Group B (Active Comparator): pursed lip breathing without Mat Pilates Training
  Interventions: Other: pursed lip breathing without Mat Pilates Training

INTERVENTIONS:
Other: Pursed lip Breathing along Mat Pilates — Experimental Group: will be treated with Pursed lip Breathing along Mat Pilates Training.
  Arms: Group A
Other: pursed lip breathing without Mat Pilates Training — Control Group will be treated pursed lip breathing without Mat Pilates Training
  Arms: Group B

SUMMARY:
Obesity is defined as BMI more than or equal to 30kg/m2. It is responsible for manifestation of serious health problem. Accumulation of adipose tissue in thorax and abdomen causes stiffness of chest, reduction in lung compliance and favoring airway closure. As result, reduction in lung volume and capacity occurs which requires increased breathing to maintain adequate oxygenation. These changes lead to limitations in activities of daily life. A Randomized Control study will be conduct to see the effects of Pilates exercise and pursed lip breathing to improve the breathing and thoracoabdominal expansion. The study will be completed within 10 months after approval of synopsis. The sample size of 34 subjects will be taken: 17 with Pilates method and 17 without Pilates method with 12% attrition rate. Pre assessment and Post assessment will be made through IPAQ questionnaire for physical activity measurement, Borg's scale (CR-10) for dyspnea measurement and Cirtometry for thoracoabdominal expansion. Study will be conducted at Star gym for women Al-Rehman Garden community, Lahore. Data will be analyzed through SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Age(25-55 years)
* Female
* Dyspnea during intense exercise 0-10
* No experience of Pilates exercise training
* BMI > 30 kg/m2

Exclusion Criteria:

* Smoking
* Pregnancy
* Practice of high intensity endurance training (squats, planks, lunges)

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Borg scale (CR-10) Questionnaire | 12 Weeks
  It is valid questionnaire and is used to measure level of Dyspnea
Thoracoabdominal expansion measurement through tape measuring tool (cirtometry). | 12 Weeks
  Thoracoabdominal expansion will be measured by means of cirtometry (tape measuring) by measuring three regions (axillary, xiphoid and abdominal).
Physical activity measurement through IPAQ questionnaire( International Physical Activity Questionnaire | 12 Weeks
  It is standardized Questionnaire to evaluate the Physical Activity of subjects. Before starting of study, the activity behavior of the participants will be monitored through IPAQ questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Star Gym for Women Al- Rehman Garden Community, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flegal KM, Carroll MD, Kuczmarski RJ, Johnson CL. Overweight and obesity in the United States: prevalence and trends, 1960-1994. Int J Obes Relat Metab Disord. 1998 Jan;22(1):39-47. doi: 10.1038/sj.ijo.0800541. PMID 9481598
- [Background] Bray GA. Medical consequences of obesity. J Clin Endocrinol Metab. 2004 Jun;89(6):2583-9. doi: 10.1210/jc.2004-0535. PMID 15181027
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Vatwani A. Pursed Lip Breathing Exercise to Reduce Shortness of Breath. Arch Phys Med Rehabil. 2019 Jan;100(1):189-190. doi: 10.1016/j.apmr.2018.05.005. Epub 2018 Jul 19. No abstract available. PMID 30033163
- [Background] Giacomini MB, da Silva AM, Weber LM, Monteiro MB. The Pilates Method increases respiratory muscle strength and performance as well as abdominal muscle thickness. J Bodyw Mov Ther. 2016 Apr;20(2):258-64. doi: 10.1016/j.jbmt.2015.11.003. Epub 2015 Nov 10. PMID 27210841
- [Background] Parisien-La Salle S, Abel Rivest E, Boucher VG, Lalande-Gauthier M, Morisset J, Manganas H, Poirier C, Comtois AS, Dube BP. Effects of Pursed Lip Breathing on Exercise Capacity and Dyspnea in Patients With Interstitial Lung Disease: A RANDOMIZED, CROSSOVER STUDY. J Cardiopulm Rehabil Prev. 2019 Mar;39(2):112-117. doi: 10.1097/HCR.0000000000000387. PMID 30624373
- [Background] Campos JL, Vancini RL, Rodrigues Zanoni G, Barbosa de Lira CA, Santos Andrade M, Jacon Sarro K. Effects of mat Pilates training and habitual physical activity on thoracoabdominal expansion during quiet and vital capacity breathing in healthy women. J Sports Med Phys Fitness. 2019 Jan;59(1):57-64. doi: 10.23736/S0022-4707.17.07908-7. Epub 2017 Oct 27. PMID 29083130